CLINICAL TRIAL: NCT01548092
Title: A Phase II Clinical Trial to Study the Feasibility and Safety of Stromal Vascular Derived From Adipose Tissue for the Treatment of Recto-vaginal Fistula
Brief Title: Stromal Vascular Fraction (SVF) for Treatment of Recto-vaginal Fistula
Acronym: HULPCIR
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC10-343; 2010-024330-35 (EudraCT Number)
Record Dates: First submitted 2012-02-26; First posted 2012-03-08 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Recto-vaginal Fistula
Keywords: Recto-vaginal fistula; Adipose Derived Stem Cells
MeSH Terms: conditions — Rectovaginal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous SVF (Experimental): Intralesional application
  Interventions: Drug: Adipose-derived stem cells without expanded

INTERVENTIONS:
Drug: Adipose-derived stem cells without expanded — Administration will be intralesional injection of cells suspension. They will be placed into fistula walls
  Other Names: Adipose-Derived Mesenchymal Stem Cells

SUMMARY:
The purpose of this study is to determine safety of Stromal Vascular Fraction (SVF) for the treatment of recto-vaginal fistula.

DETAILED DESCRIPTION:
SF-12 Test

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Recto-vaginal fistula
* Men and women over 18 years old. Good general state of health according to the findings of the clinical history and the physical examination
* Crohn's disease diagnosed at least 3 months before accepting the clinical criteria

Exclusion Criteria:

* Presence of severe proctitis or dominant active luminal disease requiring immediately therapy
* Patients with an abscess unless a complete toilet of the area with drainage of the collections and the absence of abscess and other collections is confirmed prior to treatment start
* Patients with a history of abuse of alcohol or other addictive substances in the 6 months prior to inclusion
* Patients with malignant tumor, except for basal cell or cutaneous squamous cell carcinoma, or patients with a prior history of malignant tumors, unless the neoplastic disease has been in remission for the previous 5 years
* Patients with cardiopulmonary disease which, in opinion of the investigator, in unstable or sufficiently serious to exclude the patient from the study.
* Patients with any type of medical or psychiatric disease which, in the opinion of the investigator, could be grounds for exclusion from study
* Patients with congenital or acquired immunodeficiencies. HIV, hepatitis B virus (HBV), hepatitis C virus (HCV) or treponema infection, whether active or latent
* Patients who have suffering major surgery or severe trauma in the prior 6 months
* Pregnant or breastfeeding women
* Patients currently receiving, or having received within 1 month prior to enrollment into this clinical trial, any investigational drug.
* Crohns Disease Activity Index (CDAI) Index above 200

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-07 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Safety of treatment of treated recto-vaginal fistulae. Percentage of treated enterocutaneous fistulae and percentage of subjects with closed fistulae | 16 weeks
  Safety by control the adverse effects associated with treatment Fistula close by 3D ultrasound

SECONDARY OUTCOMES:
Quality of life assessment using the SF-12 Questionnaire | 1, 4, 16, 24 weeks
  Test SF-12 of quality of life
Adverse events | 1, 4, 12, 24 weeks
  Control by investigation team of CRD (data collections)

CONTACTS AND LOCATIONS:
Overall Officials: Mariano García Arranz, PhD, Principal Investigator — Cell Therapy laboratory and general Surgery Department, Hospital Universitario La Paz
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain

REFERENCES:
- [Background] Garcia-Olmo D, Garcia-Arranz M, Garcia LG, Cuellar ES, Blanco IF, Prianes LA, Montes JA, Pinto FL, Marcos DH, Garcia-Sancho L. Autologous stem cell transplantation for treatment of rectovaginal fistula in perianal Crohn's disease: a new cell-based therapy. Int J Colorectal Dis. 2003 Sep;18(5):451-4. doi: 10.1007/s00384-003-0490-3. Epub 2003 May 20. PMID 12756590
- [Background] Garcia-Olmo D, Garcia-Arranz M, Herreros D, Pascual I, Peiro C, Rodriguez-Montes JA. A phase I clinical trial of the treatment of Crohn's fistula by adipose mesenchymal stem cell transplantation. Dis Colon Rectum. 2005 Jul;48(7):1416-23. doi: 10.1007/s10350-005-0052-6. PMID 15933795
- [Background] Herreros Marcos D, Garcia-Arranz M,Pascual Miguelañez I, Garcia-Olmo D. THE ROLE OF STEM CELLS IN SUPPURATIVE ENVIROMENTS. Experimental Dermatology 2006, 15 (6): 482
- [Background] Garcia-Olmo D, Herreros D, Pascual M, Pascual I, De-La-Quintana P, Trebol J, Garcia-Arranz M. Treatment of enterocutaneous fistula in Crohn's Disease with adipose-derived stem cells: a comparison of protocols with and without cell expansion. Int J Colorectal Dis. 2009 Jan;24(1):27-30. doi: 10.1007/s00384-008-0559-0. Epub 2008 Aug 12. PMID 18696086
- [Background] Alvarez PD, Garcia-Arranz M, Georgiev-Hristov T, Garcia-Olmo D. A new bronchoscopic treatment of tracheomediastinal fistula using autologous adipose-derived stem cells. Thorax. 2008 Apr;63(4):374-6. doi: 10.1136/thx.2007.083857. PMID 18364447
- [Background] Vilalta M, Degano IR, Bago J, Gould D, Santos M, Garcia-Arranz M, Ayats R, Fuster C, Chernajovsky Y, Garcia-Olmo D, Rubio N, Blanco J. Biodistribution, long-term survival, and safety of human adipose tissue-derived mesenchymal stem cells transplanted in nude mice by high sensitivity non-invasive bioluminescence imaging. Stem Cells Dev. 2008 Oct;17(5):993-1003. doi: 10.1089/scd.2007.0201. PMID 18537463
- [Background] Garcia-Olmo D, Herreros D, Pascual I, Pascual JA, Del-Valle E, Zorrilla J, De-La-Quintana P, Garcia-Arranz M, Pascual M. Expanded adipose-derived stem cells for the treatment of complex perianal fistula: a phase II clinical trial. Dis Colon Rectum. 2009 Jan;52(1):79-86. doi: 10.1007/DCR.0b013e3181973487. PMID 19273960
- [Background] Pascual I, de Miguel GF, Gomez-Pinedo UA, de Miguel F, Arranz MG, Garcia-Olmo D. Adipose-derived mesenchymal stem cells in biosutures do not improve healing of experimental colonic anastomoses. Br J Surg. 2008 Sep;95(9):1180-4. doi: 10.1002/bjs.6242. PMID 18690635
- [Background] García Olmo D, Trébol J, Herreros D, Garcia-Arranz M, Gonzalez M. TREATMENT OF FISTULAS USING ADIPOSE-DERIVED STEM CELLS. En: García Olmo D, García-Verdugo JM, Alemany J, Gonzalez M, Gutierrez-Fuentes JA. CELL THERAPHY . Ed. Mac Graw Hill. Madrid 2007)
- [Background] Garcia-Olmo D, Garcia-Arranz M, Herreros D. Expanded adipose-derived stem cells for the treatment of complex perianal fistula including Crohn's disease. Expert Opin Biol Ther. 2008 Sep;8(9):1417-23. doi: 10.1517/14712598.8.9.1417. PMID 18694359
- [Background] Garcia-Olmo, D; Guadalajara, H; Trebol, J, García-Arranz M. Expanded Adipose-Derived Stem Cells for the Treatment of Complex Perianal Fistula. HUMAN GENE THERAPY 2009. 20 (9):1028-1028
- [Background] Trebol, J; Garcia-Arranz, M; Georgiev-Hristov, T, et al. Cell Therapy for Enterocutaneous Fistula Associated with Crohn's Disease: A Clinical and Biological Comparison of Protocols With and Without Cell Expansion. HUMAN GENE THERAPY 2009. 20 (9): 1045-1045
- [Background] Garcia-Gomez, I; Olmedillas, S; Garcia-Arranz, M, et al. Adipose-Derived Stem Cells Reduce Abdominal Adhesion Formation in a Rat Experimental Model. HUMAN GENE THERAPY 2009. 20 (9): 1047-1047
- [Background] Georgiev-Hristov, T; Garcia-Olmo, D; Alvarez, PDA, et al. Use of Surgical Sutures Enriched with Adipose-Derived Stem Cells for Tracheal Anastomosis in Rats. HUMAN GENE THERAPY 2009. 20 (9): 1074-1075
- [Background] Vicente, A; Vazquez, MN; Entrena, A, Gqarcía-Arranz M,et al. BMP-4 Regulates the Expansion and Survival of Human Adipose Mesenchymal Cells. HUMAN GENE THERAPY .2009. 20 (9):1080-1081
- [Background] Garcia-Olmo DC, Dominguez C, Garcia-Arranz M, Anker P, Stroun M, Garcia-Verdugo JM, Garcia-Olmo D. Cell-free nucleic acids circulating in the plasma of colorectal cancer patients induce the oncogenic transformation of susceptible cultured cells. Cancer Res. 2010 Jan 15;70(2):560-7. doi: 10.1158/0008-5472.CAN-09-3513. Epub 2010 Jan 12. PMID 20068178
- [Background] Garcia-Arranz M, Gomez-Pinedo U, Hardisson D, Herreros D, Guadalajara H, Garcia-Gomez I, Garcia-Verdugo JM, Garcia-Olmo D. Histopathological analysis of human specimens removed from the injection area of expanded adipose-derived stem cells. Histopathology. 2010 Jun;56(7):979-82. doi: 10.1111/j.1365-2559.2010.03573.x. No abstract available. PMID 20636801
- [Background] Tihomir Georgiev-Hristov, M.D.; Ignacio García-Gómez, Ph.D.; Prudencio Díaz-Agero, M.D.; Luz Vega-Clemente; Jacobo Trébol, M.D.; Damián García-Olmo, M.D., Ph.D.; Mariano García-Arranz, Ph.D. "SUTURES ENRICHED WITH ADIPOSE-DERIVED STEM CELLS FOR ENHANCED HEALING OF TRACHEAL ANASTOMOSIS IN RATS" Histology and Histopathology. 2010 (UNDER REVISION)
- [Background] Garcia-Olmo D, Herreros D, De-La-Quintana P, Guadalajara H, Trebol J, Georgiev-Hristov T, Garcia-Arranz M. Adipose-derived stem cells in Crohn's rectovaginal fistula. Case Rep Med. 2010;2010:961758. doi: 10.1155/2010/961758. Epub 2010 Mar 7. PMID 20224798
- [Background] Pascual I, De Miguel Fernandez G, García-Arranz M, García-Olmo D.